CLINICAL TRIAL: NCT00534287
Title: Prospective, Randomized, Open, Multicentre Study About the Effect of an Empirical Antibiotic Monotherapy With Meropenem (Meronem®) Versus a Combination Therapy With Moxifloxacin (Avalox®) on Organ Dysfunction in Patients With Severe Sepsis and Septic Shock
Brief Title: Comparison of Two Antibiotic Regimen (Meropenem Versus Meropenem+Moxifloxacin)in the Treatment of Severe Sepsis and Septic Shock
Acronym: MaxSep
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kompetenznetz Sepsis (Network)
Collaborators: AstraZeneca (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2006-006984-21; bmbf grant: 01 KI 01 06
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: sepsis; antibiotics; carbapenems; fluoroquinolones; Severe sepsis and septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Meropenem; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MeroMono (Active Comparator): Monotherapy with meropenem
  Interventions: Drug: meropenem
- MeroMoxi (Active Comparator): Combination therapy with meropenem + moxifloxacin
  Interventions: Drug: meropenem, moxifloxacin

INTERVENTIONS:
Drug: meropenem — Empirical antibiotic therapy with 3 x 1 g intravenous meropenem. Dosage is adjusted in case of renal dysfunction. Recommended duration of therapy is 7 days but can be extended up to 14 days.
  Other Names: Meronem® (meropenem)
  Arms: MeroMono
Drug: meropenem, moxifloxacin — Empirical antibiotic therapy with 3 x 1 g intravenous meropenem plus 1 x 400 mg intravenous moxifloxacin. Dosage of meropenem is adjusted in case of renal dysfunction. Recommended duration of therapy is 7 days but can be extended up to 14 days.
  Other Names: Meronem® (meropenem); Avalox® (moxifloxacin)
  Arms: MeroMoxi

SUMMARY:
Severe sepsis and septic shock are diseases of infectious origin with a high risk of death. Antibiotic therapy is mandatory but it is unknown whether one antibiotic alone is sufficient for initial therapy. The purpose of this study is to compare a therapy with meropenem alone or the combination of meropenem plus moxifloxacin in the treatment of severe sepsis/ septic shock. Patients randomly receive one of the two treatments for at least 7 days but not longer than 14 days.

DETAILED DESCRIPTION:
Early intravenous empiric broad-spectrum antimicrobial therapy is an essential part of sepsis therapy. Inadequacy of empirical antibiotic therapy is associated with an increased mortality rate. Carbapenems are designed for empirical antimicrobial monotherapy. Combination therapy has been suggested but efficiency remains to be proven. In this study, antimicrobial monotherapy with meropenem is compared with a combination therapy of meropenem and moxifloxacin. It is hypothesized that the superior antibiotic therapy is associated with a lower overall organ dysfunction in sepsis. Study therapy lasts for at least 7 days unless microbiological results suggest otherwise. Study therapy may be extended to 14 days. Follow up examinations occur at 28 and 90 days. This investigator initiated study is supported by the German government (bmbf) and unrestricted industrial grants.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis or septic shock according to ACCP/SCCM criteria
* Onset of severe sepsis or septic shock <24 h
* Informed consent
* Effective contraception in fertile women

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Breast-feeding women
* Pretreatment with meropenem, imipenem, or ertapenem within the last 4 weeks (>1 daily dosage)
* Pretreatment with moxifloxacin,ciprofloxacin, or levofloxacin within the last 4 weeks (>1 daily dosage)
* Pretreatment with a pseudomonas effective cephalosporin (cefepime, ceftazidim, cefpirom) or piperacillin within the last 48 hours (>1 daily dosage).
* Pretreatment with other chinolones within the last 4 weeks (>1 daily dosage)
* Presence of infection where guidelines recommend another antimicrobial therapy than the study medication (i.e. endocarditis)
* Evidence or strong clinical suspicion of a microorganism where the study medication is known to be ineffective (i.e. tuberculosis, MRSA- or VRE-infection)
* Known allergy against meropenem or moxifloxacin
* Tendon disease or injury due to past quinolone therapy
* Congenital or acquired prolongation of QT-interval
* Concomitant medication which prolongs the QT-interval
* Electrolyte imbalance, especially uncorrected hypokalemia
* Clinically relevant bradycardia
* Clinically relevant cardiac dysfunction with reduced left-ventricular ejection fraction
* Symptomatic arrhythmias in the medical history
* Significant hepatic impairment (Child-Pugh C) or elevation of liver enzymes >5x the upper normal range
* No commitment to full patient support (i.e. DNR order)
* Patient's death is considered imminent due to coexisting disease
* Concomitant participation in another study or study participation with in the last 30 days.
* Relationship of the patient to study team member (i.e. colleague, relative)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2007-10; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Mean total SOFA score | study duration but not longer than 14 days

SECONDARY OUTCOMES:
Mortality | 28 and 90 days
ICU and hospital length of stay
Response to therapy | day 7 and day 10
Clinical and microbiological cure | End of study therapy (day 7-14) and release from ICU (max. day 21)
Frequency of adverse events (AEs, SAEs, SUSARs)
Ventilator free days | 28 and 90 days
Days without renal replacement therapy | 28 and 90 days
Vasopressor free days | 28 and 90 days
SOFA-subscores
Antibiotics free days | 28 and 90 days
Costs of antibiotic therapy | ICU stay
Frequency of resistances to antibiotics | ICU stay
Frequency of new infections

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Reinhart, MD, Study Chair — University Hospital Jena; Dep. of Anesthesiology and Intensive Care Medicine; Markus Löffler, MD, Study Director — University Leipzig; Koordinierungszentrum für Klinische Studien Leipzig (KKSL); Thomas Deufel, MD, Study Director — University Hopitel Jena, Institute for Medical Chemistry
Locations (52):
- Germany (52):
  - University Hospital Aachen - Dep. of Anesthesiology, Aachen
  - Klinikum Augsburg - Dep. of Anesthesiology and Intensive Care Medicine, Augsburg
  - Charité Berlin - Dep. of Anesthesiology and Intensive Care Medicine, Berlin
  - Charité Berlin - Dep. of Medicine (Cardiology, Angiology, Pneumology), Berlin
  - Charité Campus Mitte -Dep.of Infectiology and Pneumonology, Berlin
  - Charité Campus Benjamin Franklin - Dep. of Medicine IV, Berlin
  - Vivantes Klinikum Neukölln - Cardiology, Berlin
  - Vivantes Klinikum Neukölln - Dep. of Anesthesiology, Intensive Care Medicine and Pain Therapy, Berlin
  - Charité Berlin - Campus Virchow-Klinikum - Dep. of Nephrology, Berlin
  - Ev. Krankenhaus Gilead I - Dep. of Anesthesiology and Intensive Care Medicine, Bielefeld
  - University Hospital Bonn - Dep. of Anesthesiology and Intensive Care Medicine, Bonn
  - Städtisches Klinikum Brandenburg - Intensive Care Unit, Brandenburg
  - University Hospital Köln - Dep. of Internal Medicine I, Cologne
  - Hospital Merheim - Dep. of Anesthesiology and Intensive Care Medicine, Cologne
  - Klinikum Darmstadt - Dep. of Anesthesiology, Intensive Care Medicine and Pain Therapy, Darmstadt
  - Klinikum Dessau - Dep. of Medicine, Dessau
  - Hospital Lippe-Detmold - Dep. of Anesthesiology and Intensive Care Medicine, Detmold
  - Krankenhaus Dresden-Friedrichstadt, Dresden
  - University Hospital Dresden - Dep. of Anesthesiology and Intensive Care Med., Dresden
  - HELIOS Klinikum Erfurt - Dep. of Anesthesiology and Intensive Care Medicine, Erfurt
  - University Erlangen-Nürnberg - Dep. of Medicine IV, Erlangen
  - University Hospital Freiburg - Dep. of Medicine III, Freiburg im Breisgau
  - Klinik am Eichert - Dep. of Anesthesiology, Intensive Care Medicine, and Pain Therapy, Göppingen
  - Georg August Universität Göttingen - Dep. of Anesthesiology and Intensive Care Medicine, Göttingen
  - Ernst-Moritz-Arndt-Universität Greifswald - Dep. of Anesthesiology and Intensive Care Medicine, Greifswald
  - Ernst-Moritz-Arndt-Universität Greifswald, Dep. of Internal Medicine B, Greifswald
  - Martin-Luther-Universität Halle-Wittenberg - Dep. of Anesthesiology and Intensive Care Medicine, Halle
  - Hospital Martha-Maria Halle-Dölau gGmbH - Dep. of Anesthesiology and Intensive Care Medicine, Halle
  - Universitätsklinikum Hamburg-Eppendorf - Dep. of Intensive Care Medicine, Hamburg
  - Klinikum Hannover Nordstadt - Dep. of Anesthesiology and Intensive Care Medicine, Hanover
  - Medizinische Hochschule Hannover, Dep. of Internal Medicine/ Pneumology, Hanover
  - Westküstenklinikum Heide - Dep. of Anesthesiology and Intensive Care Medicine, Heide
  - University Hospital Heidelberg - Dep. of Medicine IV, Heidelberg
  - University Hospital Heidelberg - Dep. of Visceral and Transplantation Surgery, Heidelberg
  - University Hospital Saarland - Deop. of Anesthesiology, Intensive Care Medicine, and Pain Therapy, Homburg/Saar
  - University Hospital Jena, Dep. of Anesthesiology and Intensive Care Medicine, Jena
  - University Hospital Kiel - Dep. of. Anesthesiology and Intensive Care Medicine, Kiel
  - University Hospital Leipzig - Dep. of Anesthesiology and Intensive Care Medicine, Leipzig
  - Hospital Ludwigshafen am Rhein - Dep. of Cardiac Surgery, Ludwigshafen
  - Klinikum Lüdenscheid - Dep. of Anesthesiology, Lüdenscheid
  - University Hospital Mannheim - Dep. of Medicine I, Mannheim
  - University Hospital Munich - Dep. of Internal Medicine, Munich
  - Hospital Munich Harlaching - Dep. of Internal Acute Medicine and Prevention, Munich
  - Klinikum rechts der Isar - Dep. of Anesthesiology, Munich
  - University Hospital Münster - Dep. of Anesthesiology and Intensive Care Medicine, Münster
  - Klinikum Oldenburg - Dep. of Anesthesiology, Intensive Care Medicine, Emergency Medicine, Pain Therapy, Oldenburg
  - Klinikum Ernst von Bergmann - Dep. of Anesthesiology and Intensive Care Medicine, Potsdam
  - University Hospital Rostock - Dep. of Anesthesiology and Intensive Care Medicine, Rostock
  - Ev. Jung-Stilling-Krankenhaus - Dep. of Anesthesiology, Intensive Care Medicine, Emergency Medicine, Siegen
  - University Hospital Tübingen - Dep. of Medicine, Tübingen
  - University Hospital Ulm - Dep. of Internal Medicine II, Ulm
  - Stiftung Juliusspital Würzburg - Dep. of Medicine (Cardiology), Würzburg

REFERENCES:
- [Background] American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference: definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. Crit Care Med. 1992 Jun;20(6):864-74. PMID 1597042
- [Background] Reinhart K, Brunkhorst F, Bone H, Gerlach H, Grundling M, Kreymann G, Kujath P, Marggraf G, Mayer K, Meier-Hellmann A, Peckelsen C, Putensen C, Quintel M, Ragaller M, Rossaint R, Stuber F, Weiler N, Welte T, Werdan K; Deutsche Sepsis-Gesellschaft e.V. [Diagnosis and therapy of sepsis: guidelines of the German Sepsis Society Inc. and the German Interdisciplinary Society for Intensive and Emergency Medicine]. Anaesthesist. 2006 Jun;55 Suppl 1:43-56. German. PMID 17051663
- [Background] Bochud PY, Bonten M, Marchetti O, Calandra T. Antimicrobial therapy for patients with severe sepsis and septic shock: an evidence-based review. Crit Care Med. 2004 Nov;32(11 Suppl):S495-512. doi: 10.1097/01.ccm.0000143118.41100.14. PMID 15542958
- [Background] Harbarth S, Garbino J, Pugin J, Romand JA, Lew D, Pittet D. Inappropriate initial antimicrobial therapy and its effect on survival in a clinical trial of immunomodulating therapy for severe sepsis. Am J Med. 2003 Nov;115(7):529-35. doi: 10.1016/j.amjmed.2003.07.005. PMID 14599631
- [Background] Safdar N, Handelsman J, Maki DG. Does combination antimicrobial therapy reduce mortality in Gram-negative bacteraemia? A meta-analysis. Lancet Infect Dis. 2004 Aug;4(8):519-27. doi: 10.1016/S1473-3099(04)01108-9. PMID 15288826
- [Background] Engel C, Brunkhorst FM, Bone HG, Brunkhorst R, Gerlach H, Grond S, Gruendling M, Huhle G, Jaschinski U, John S, Mayer K, Oppert M, Olthoff D, Quintel M, Ragaller M, Rossaint R, Stuber F, Weiler N, Welte T, Bogatsch H, Hartog C, Loeffler M, Reinhart K. Epidemiology of sepsis in Germany: results from a national prospective multicenter study. Intensive Care Med. 2007 Apr;33(4):606-18. doi: 10.1007/s00134-006-0517-7. Epub 2007 Feb 24. PMID 17323051
- [Background] Pletz MW, Bloos F, Burkhardt O, Brunkhorst FM, Bode-Boger SM, Martens-Lobenhoffer J, Greer MW, Stass H, Welte T. Pharmacokinetics of moxifloxacin in patients with severe sepsis or septic shock. Intensive Care Med. 2010 Jun;36(6):979-83. doi: 10.1007/s00134-010-1864-y. Epub 2010 Mar 25. PMID 20336279
- [Result] Brunkhorst FM, Oppert M, Marx G, Bloos F, Ludewig K, Putensen C, Nierhaus A, Jaschinski U, Meier-Hellmann A, Weyland A, Grundling M, Moerer O, Riessen R, Seibel A, Ragaller M, Buchler MW, John S, Bach F, Spies C, Reill L, Fritz H, Kiehntopf M, Kuhnt E, Bogatsch H, Engel C, Loeffler M, Kollef MH, Reinhart K, Welte T; German Study Group Competence Network Sepsis (SepNet). Effect of empirical treatment with moxifloxacin and meropenem vs meropenem on sepsis-related organ dysfunction in patients with severe sepsis: a randomized trial. JAMA. 2012 Jun 13;307(22):2390-9. doi: 10.1001/jama.2012.5833. PMID 22692171
- See also: Competence Network Sepsis (SepNet) — http://www.sepsis-gesellschaft.de/DSG/Deutsch/SepNet?sid=nbGlH39rI6b9u2fBVVhxiM&iid=1
- See also: German Sepsis Society — http://www.sepsis-gesellschaft.de/